CLINICAL TRIAL: NCT05791682
Title: "Comparative Clinical Evaluation of Microfilled Resin Sealant, Nanofilled Resin Sealant and Flowable Composite as Sealant With Unfilled Resin Sealant on Permanent First Molar Teeth in Children."
Brief Title: "Comparative Clinical Evaluation of Pit and Fissure Sealants on Permanent First Molar Teeth in Children."
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PGIDS/BHRC/21/14
Record Dates: First submitted 2022-11-12; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: PITS AND FISSURE SEALANT
MeSH Terms: interventions — Pit and Fissure Sealants

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MICROFILLED RESIN SEALANT (Active Comparator): -Microfilled rein sealant (fissurit FX) after etching, washing, drying, sealant was gradually applied along the fissure of first permanent molar, Immediately light cured for 20 sec
  Interventions: Drug: Sealant, Fissure
- NANOFILLED RESIN SEALANT (Active Comparator): Nanofilled resin sealant (Grandioseal) after etching, washing, drying, sealant was gradually applied along the fissure. Immediately light cured for 20 sec.
  Interventions: Drug: Sealant, Fissure
- FLOWABLE COMPOSITE (Active Comparator): Flowable composite (Te-Econom Flow) after etching, washing, drying, adhesive was applied and dried under gentle air flow for 2-3 sec and was light cured. A uniform layer of flowable composite was applied and light cure for 20 sec.
  Interventions: Drug: Sealant, Fissure
- UNFILLED RESIN SEALANT (Active Comparator): Unfilled resin sealant (clinpro) after etching, washing, drying, sealant will be gradually applied along the fissure. Immediately light cure for 20 sec.
  Interventions: Drug: Sealant, Fissure

INTERVENTIONS:
Drug: Sealant, Fissure — FISSURIT FX- MICROFILLED RESIN SEALANT WITH 55% FILLER GRANDIOSEAL- NANOFILLED RESIN SEALANT WITH 70% FILLER TE-ECONOM- FLOW -FLOWABLE COMPOSITE AS SEALANT CLINPRO TM- UNFILLED RESIN SEALANT

SUMMARY:
Study was aimed to evaluate and compare clinical efficacy of the Microfilled resin sealant, Nanofilled resin sealant, Flowable composite as sealant, with Unfilled resin sealant on first permanent molar in children at 9 months follow ups.

Children (age 7 to 10) with deep pits and fissures, (ICDAS 0-2) included in the study and study was Split mouth randomized controlled clinical trial.

Sample size- Total number of 42 patients will be recruited in the study, with 42 first permanent molars in each group.

Methods-Patients were seated in supine position on the dental chair and cotton rolls will be applied for isolation. The first permanent molar in each group was treated as follows:

Group 1 -Intervention with Microfilled resin sealant. Group 2- ¬Intervention with Nanofilled resin sealant. Group 3 -Intervention with Flowable composite as sealant. Group 4 - ¬Intervention with Unfilled resin sealant. Patients and their parents were received instructions for daily brushing and oral hygiene maintenance. Sealant clinical efficacy was evaluated at 3, 6 and 9 month recall visit.

OUTCOME MEASURES:

1. Primary outcomes: To evaluate sealant retention, anticaries effect and marginal integration.
2. Secondary outcomes: to evaluate, colour change and surface roughness of sealant.

ELIGIBILITY:
Inclusion crieteria

1. Normal healthy children aged 7 to 10 years.
2. Subjects who are not undergoing any other preventive dental health treatment.
3. Availability for the duration of the study.
4. Satisfactory dental care performed at home.
5. The willingness of the patient to accept the treatment.
6. All four first permanent molars that have completely erupted with deep pits and fissures.
7. Fissures either intact, sound or retentive which are stained, caries free or ICDAS 0-2.

EXCLUSION CRITERIA

1. Children whose parents will not give informed consent.
2. Special child, a child with compromised systemic health.
3. Long-term medication affecting the salivary flow.
4. Children enrolled for other studies or fluoridation program.
5. Adverse reaction reported to any dental material.
6. Uncooperative child.
7. Bruxism or malocclusion.
8. Children with developmental defects/ hypoplastic molars or caries affected teeth (ICDAS>2).
9. Teeth with restoration and partially retained sealants.
10. Children who cannot come for the follow-up.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
To evaluate sealant retention | 9 months
  Alpha - complete retention Bravo- partial retention Charlie- no retention

SECONDARY OUTCOMES:
To evaluate marginal integrity | 9 months
  Alpha- No visible evidence of a crevice along the margin of the sealant that the explorer could penetrate.
  Bravo- Visible evidence of a crevice along the margin of the sealant that the explorer could penetrate.
to evaluate anti caries effect | 9 months
  Alpha- Sound fissures. Bravo- Fissures with caries.
to evaluate colour change | 9 months
  Alpha- No discoloration anywhere on the margin around the sealant. Bravo- Visible partial discoloration the margin around sealant. Charlie- Visible discoloration on the margin around all sealant.
to evaluate surface roughness | 9 months
  Alpha- The sealant is similar to polished enamel. Bravo- The sealant surface is similar to composite material surface contained submicron filler.
  Charlie- The surface is rough that prevents the explorer movement along the surface.

CONTACTS AND LOCATIONS:
Locations (1):
- Post graduate institute of dental sciences, Rohtak, Haryana, India